CLINICAL TRIAL: NCT03404622
Title: : Immediate Post-placental Insertion of the Intrauterine Contraceptive Device During Cesarean Delivery Versus 6 Week Post-Cesarean Insertion
Brief Title: Immediate Post-placental Insertion of IUCD During Cesarean Delivery Versus 6 Week Post-Cesarean Insertion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ALshaimaa Aboalhassan Ali (Other)
Responsible Party: Sponsor-Investigator, ALshaimaa Aboalhassan Ali, physician, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: shom
Record Dates: First submitted 2018-01-10; First posted 2018-01-19 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Mechanical Complication of Intrauterine Device

STUDY DESIGN:
Intervention Model Description: 200 pregnant women will be included in this study, will be divided into two groups Group 1 IUCD will be inserted immediate post-placental removal and include 100 pregnant women Group2 IUCD will be inserted 6 weeks postpartum and include 100 pregnant women.
Who Masked: Participant, Care Provider
Masking Description: Randomization will be based on the sequence generation created by computer and randomization tablets. Consenting patients fulfilling inclusion criteria will be randomizes into one of the following 2 groups. Randomized allocation will be kept in opaque sealed envelopes, with enrollment numbers written on the envelopes. the envelopes will contain a card on with the designated study group will be written. after enrollment of the patients in the study , the envelopes marked with study number will be unsealed and the patients allocated to either groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Postplacental IUCD Insertion during Cesarean section (Active Comparator): IUCD inserted postplacental removal
  Interventions: Drug: IUCD
- 6 Week Post-Cesarean Insertion of IUCD (Active Comparator): IUCD inserted after six weeks post Cesarean section delivery
  Interventions: Drug: IUCD

INTERVENTIONS:
Drug: IUCD — IUCD will be inserted in 100 women post placental removal and will be inserted in anther 100 women after six weeks post cesarean delivery

SUMMARY:
The aim of current study is to compare the rates of IUCD expulsion and complications in immediate post-placental insertion versus delayed IUCD insertion (6-weeks after cesarean delivery)

DETAILED DESCRIPTION:
Intrauterine devices (IUDs) are among the most effective forms of contraception, offering greater than 99% efficacy per year of use and are completely reversible .

Post-placental intrauterine device (IUD) insertion is a safe, convenient, and effective option for postpartum contraception. "Post-placental" refers to insertion within 10-15 minutes of placental delivery, after vaginal or cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 -45
* Singleton pregnancy at ≥32 weeks gestation at time of enrollment
* Voluntarily requesting to IUD placement for postpartum contraception
* Able to give consent and agree to the terms of the study

Exclusion Criteria:

1. Uterine anomaly that preventing replacement of IUD.
2. Chorioamnionitis (such as prolonged rupture of membranes >18 hours, prolonged labor >24 hours, fever >38C).
3. Puerperal sepsis and unresolved postpartum hemorrhage.
4. IUD allergy (copper).
5. Systemic lupus erythematosus with severe thrombocytopenia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 200 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Expulsion | 3 months
  The time until expulsion of the IUD will be defined as the time from insertion until expulsion occurred, if known. If the date of expulsion is not known, this will be documented as the day after the IUD was last known to be in place. If a pregnancy is detected and the IUD is absent (and the participant was unaware of expulsion), the expulsion will be assumed to have occurred at the time of conception, as determined by gestational age on ultrasound. Expulsions will be measured as total expulsions and separately noted whether complete or partial

SECONDARY OUTCOMES:
Displacement | 3 months
  The displacement is diagnosed by doing trans-vaginal ultrasound that showed IUCD that displaced up or down word
Infection | 3 months
  The diagnosis of PID will be made based on the 2006 CDC guidelines and the criteria used in the PEACH study.
Bleeding | 3 months
  Irregular bleeding (including spotting, light bleeding, heavy or longer menstrual period) are common in the first 3 months and may persist.
Perforation | 3 months
  The diagnosis of a perforation may be made by a transvaginal sonogram that shows no IUD within the uterus and an abdominal radiograph that show IUD within the abdominal cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser M Aboutalib, MD, Study Director — Ain Shams University; Ahmed S AbdelHamid, MD, Study Director — Ain Shams University; ALshaimaa A Ali, MBBch, Principal Investigator — Ain Shams University; Haitham Torky, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sothornwit J, Kaewrudee S, Lumbiganon P, Pattanittum P, Averbach SH. Immediate versus delayed postpartum insertion of contraceptive implant and IUD for contraception. Cochrane Database Syst Rev. 2022 Oct 27;10(10):CD011913. doi: 10.1002/14651858.CD011913.pub3. PMID 36302159